CLINICAL TRIAL: NCT01627743
Title: CorRELation Between PatIent PErception of the Ability to Perform Morning Activities and Findings on Clinical Examination in COPD Patients
Brief Title: CorRELation Between PatIent PErception and Findings on Clinical Examination
Acronym: RELIEF
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RRO-ATC-2012/1
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: CDLM; visual scale - physician evaluation; COPD; GOLD group C and D
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- COPD patients grade C and D

SUMMARY:
This is a multi-center, prospective, non-interventional study that aims to evaluate in daily clinical practice, the possible corelation between patIent perception of the ability to perform morning activities and physician evaluation; patients with COPD, grade C and D.

DETAILED DESCRIPTION:
CorRELation between PatIent PErception of the Ability to Perform Morning Activities and Findings on Clinical Examination in COPD Patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD, grade C and D according to GOLD Guidelines Revised 2011
* Current or past smokers, of at least 10 pack years
* Receive any inhaled combination therapy for COPD (inhaled corticosteroid / long acting β2-agonist bronchodilator) initiated for at least one month before entering in the study

Exclusion Criteria:

* History of exacerbation of COPD symptoms within the last month before visit 1, inclusive; history of asthma or allergic rhinitis; history of lung carcinoma or any other respiratory condition that may limit the airflow circulation
* Inability to understand study procedures and inability/refuse to complete CDLM questionnaires and/or record the values showed on the pedometer screen

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients, group C and D according to GOLD guidelines 2011, being treated for at least 1 month with combination ICS/LABA treatment
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Capacity of Daily Living during the Morning (CDLM) Questionnaire | Baseline and 3 months
  CDLM questionnaire is a simple self-reporting tool of the burden and ability of COPD patients to perform routine morning activities: washing, dressing, eating breakfast, walking around. For each of these morning activities the score is varying from 0 (indicating worst case) to 5 (indicating best case).
Change from baseline of patient's general health status based upon physician evaluation - visual scale | Baseline and 3 months
  General health status visual scale is assessing the physicians perception of the patient health status following the clinical examination. Based upon clinical evaluation, the physician will indicate the patient's general condition on a a scale consisting of 5 levels. The scale will be completed at each visit and the score can vary from 1(very bad general health status) to 5 (very good general health status) .

SECONDARY OUTCOMES:
Demographic patient characteristics | Day 0 (visit1)
  Demographic patient characteristics are:
  Age (years), gender (male/female), weight (kg), height (cm), place of origin (urban, rural)
Patient adherence to treatment - visual scale | up to 3 months
  The physician will evaluate adherence to treatment, after discussion with patient, by completing a visual scale for evaluation patient's adherence to treatment (adherence will be assessed in percentage, by indicating at the scale the value from 0% to 100% adherence).
  The visual scale has the following cut-off points: 0% (no adherence to treatment), 25% (poor adherence), 50% (medium adherence), 75% (good adherence), 100% (high adherence).
Number of daily walking steps (using pedometer) | up to 3 months
  The pedometers register the total daily walking steps. Each morning, the subject will reset the device by pressing the on/reset button. At the end of the day, the patient will record the number of daily walking steps. The estimated value for number of walking steps is 2,500 - 4,500 steps/day (based on previous studies).
Number of exacerbations | up to 3 months
  Exacerbation is defined as a worsening of COPD symptoms that is beyond day-to-day variations and that requires antibiotic treatment and/or short systemic corticoid treatment and/or emergency room visit with or without hospital admission (according to GOLD criteria and previous studies).

CONTACTS AND LOCATIONS:
Overall Officials: Florin Mihaltan, PROFESSOR, Principal Investigator — University of Medicine and Pharmacy Carol Davila, Bucharest, Romania
Locations (19):
- Romania (19):
  - Research Site, Bacau
  - Research Site, Botoșani
  - Research Site, Bucharest
  - Research Site, Buzău
  - Research Site, Călăraşi
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Craiova
  - Research Site, Drobeta-Turnu Severin
  - Research Site, Fălticeni
  - Research Site, Focşani
  - Research Site, Iași
  - Research Site, Leordeni
  - Research Site, Luduş
  - Research Site, Oradea
  - Research Site, Ploieşti
  - Research Site, Râmnicu Vâlcea
  - Research Site, Reghin
  - Research Site, Slatina